CLINICAL TRIAL: NCT02944097
Title: Study of the Oral Bioavailability of Trans-epsilon-viniferin and Trans-resveratrol From Native and Micellar Solubilized vineatrol30 Vine Extract
Brief Title: Bioavailability of Resveratrol From Vineatrol30 Extract Incorporated Into Micelles
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HS-VM-2015
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Safety After Oral Intake; Pharmacokinetics After Oral Intake
Keywords: Bioavailability; Pharmacokinetics; trans-resveratrol; trans-epsilon-viniferin; Vineatrol 30

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vineatrol30 native powder (Experimental): 500 mg Vineatrol30 containing 30 mg trans-resveratrol and 75.2 mg trans-epsilon-viniferin
  Interventions: Dietary Supplement: Vineatrol 30 native powder
- Vineatrol30 micelles (Experimental): 500 mg Vineatrol30 micelles containing 30 mg trans-resveratrol and 75.2 mg trans-epsilon-viniferin
  Interventions: Dietary Supplement: Vineatrol 30 micelles

INTERVENTIONS:
Dietary Supplement: Vineatrol 30 native powder
  Arms: Vineatrol30 native powder
Dietary Supplement: Vineatrol 30 micelles
  Arms: Vineatrol30 micelles

SUMMARY:
To enhance the oral bioavailability of the antioxidants trans-resveratrol and trans-ε-viniferin from Vineatrol30 grapevine-shoot extract, the native powder was incorporated into micelles. A single dose, single blind, two arms crossover trial was conducted. Plasma and urine samples were collected at intervals up to 24 h after oral intake of native or micellar Vineatrol30 (500 mg), and resveratrol content was quantified and compared between formulations. Tolerability of the dose was also controlled by safety parameters in plasma.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers with blood chemistry values within normal ranges

Age: 18-35 years

BMI: 19-25 kg/m2

Exclusion Criteria:

Pregnancy or lactation

Alcohol and/or drug abuse

Use of dietary supplements or any medications, except contraceptives

Any known malignant, metabolic and endocrine diseases

Previous cardiac infarction

Dementia

Participation in a clinical trial within the past 6 weeks prior to recruitment

Smoking

Physical activity of more than 5 h/wk

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of plasma concentration vs. time of total trans-resveratrol [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Mean area under the curve (AUC) of plasma concentration vs. time of total trans-epsilon-viniferin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total trans-resveratrol [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total trans-epsilon-viniferin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total trans-resveratrol [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total trans-epsilon-viniferin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total trans-resveratrol [nmol/g creatinine] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total trans-epsilon-viniferin [nmol/g creatinine] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | 0, 4, 24h post-dose
Serum alanine transaminase activity [U/L] | 0, 4, 24h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 0, 4, 24h post-dose
Serum alkaline phosphatase activity [U/L] | 0, 4, 24h post-dose
Serum bilirubin | 0, 4, 24h post-dose
Serum uric acid [mg/dL] | 0, 4, 24h post-dose
Serum creatinine [mg/dL] | 0, 4, 24h post-dose
Serum total cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum HDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum LDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum triacylglycerols [mg/dL] | 0, 4, 24h post-dose
LDL/HDL cholesterol ratio | 0, 4, 24h post-dose
Serum cystatin C [mg/mL] | 0, 4, 24h post-dose
Glomerular filtration rate [mL/min] | 0, 4, 24h post-dose
Serum glucose [mg/dL] | 0, 24h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Prof. Dr, Principal Investigator — University of Hohenheim
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Website of the research group — http://www.nutrition-research.de/